CLINICAL TRIAL: NCT02276846
Title: Palpitate-Eluting Balloon Angioplasty in the Treatment of Coronary Bifurcation Lesion Evaluated by OCT
Acronym: PEBCBLO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Liu Bin, M.D.Professor Director of Cardiology Department, Second Hospital of Jilin University
Other Study IDs: SecondJilinU
Record Dates: First submitted 2014-10-12; First posted 2014-10-28 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Angioplasty; Percutaneous Coronary Intervention
Keywords: Palpitate-Eluting Balloon; Bifurcation; OCT; Transluminal

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Paclitaxel-Eluting Balloon

SUMMARY:
The aim of the study is to use optical coherence tomography (OCT) to investigate the efficacy of Paclitaxel-eluting PTCA-balloon dilation (SeQuent Please) in SB and drug eluting stent (EXCEL stent) deployment in the main branch (reference diameter: ≥ 2.5 mm and ≤ 4.0 mm, reference diameter of side branch: ≥ 2.0 mm and ≤ 3.5 mm, length of stenoses in either branch ≤ 30 mm) in the treatment of significant (>70%) de-novo-bifurcation stenoses of any Medina classification type in the native coronary artery as reflected by procedural success and to evaluate the preservation of vessel patency.

DETAILED DESCRIPTION:
Catheter interventions of coronary lesions involve a bifurcation in 15-20%. The treatment of bifurcation lesions is usually more difficult as compared to non-bifurcation lesions and the complication rate is higher. Possible complications are acute SB closure (BBC one) and higher rates of restenosis and stent thrombosis. Carina shifting after stenting ,double or triple layers of stents, stent distortion and different tissue distribution may be the reasons. The use of drug-eluding stents in the treatment of bifurcation lesions suggests that DES reduces the rate of restenosis int he main branch (5-10%); however, results in the side branch are not optimal. Current interventional treatment of most bifurcation lesions consists in implanting a DES in the MB with POBA and provisional T-stenting of the SB. Drug eluting Balloon is the new options and improvements in the field of coronary angioplasty. Clinically proven, it offers completely new procedural options to treat vascular stenoses since the drug elution does not require a stent platform. Since the SB is rarely stented, the DEB could be particularly helpful to reduce the restenosis rate of a SB lesion. PEPCAD V trial has proved Percutaneous treatment of bifurcation lesions with a drug-eluting balloon resulted in a procedural success of 100%. Follow-up angiography at nine months showed DES-like results in MB and SB. In PEPCAD V trial，the MB was dilated with a DEB. Next, a BMS (CoroflexR, B. Braun Melsungen AG, Germany) was implanted in the MB. While the procedure is complex, whether we can put drug eluting stent in MB directly and this overlap of drug delivery is harmful. OCT system had an axial resolution of 20 microm and a transverse resolution of 30 microm. OCT was able to penetrate and image near-occlusive coronary plaques. Therefore, it is prudent to use OCT to investigate the efficacy of Paclitaxel-eluting PTCA-balloon dilation (SeQuent Please) in SB and drug eluting stent (EXCEL stent) deployment in the main branch (reference diameter: ≥ 2.5 mm and ≤ 4.0 mm, reference diameter of side branch: ≥ 2.0 mm and ≤ 3.5 mm, length of stenoses in either branch ≤ 30 mm) in the treatment of significant (>70%) de-novo-bifurcation stenoses of any Medina classification type in the native coronary artery as reflected by procedural success and to evaluate the preservation of vessel patency.

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria

* Inclusion Criteria: Patient Related
* Patients with stable angina pectoris (CCS class 1-3) or with unstable angina pectoris (Braunwald class 1-2, A-C) or documented ischemia or with documented silent ischemia
* Patients eligible for coronary revascularization by means of PCI
* Patients must be 18 years of age
* Women of childbearing potential may not be pregnant nor have the desire to becoming pregnant during the first year following the study procedure. Hence, patients will be advised to use an adequate birth control method up to and including 6-month follow-up
* Patients who are mentally and linguistically able to understand the aim of the study and to show sufficient compliance in following the study protocol
* Patients must agree to undergo the 9-month angiographic follow-up
* Patients must agree to undergo the 3-year clinical follow-up
* Patient is able to verbally acknowledge and understand the associated risks, benefits, and treatment alternatives of this trial. The patients, by providing their informed consent, must agree to these risks and benefits as stated in the patient informed consent document.

Inclusion Criteria: Lesion Related

* De-novo bifurcational native left coronary artery lesion (reference diameter LAD or LCx:2.5 mm-4.0 mm, length of stenosis: ≤30 mm, reference diameter D1/D2 or OMS1/OMS2:2.0 mm -3.5 mm, length of stenosis: ≤30 mm)
* Diameter stenosis pre procedure must be either 70 % in either one or both branches of the lesion (i.e. bifurcational lesion of any type of the Medina classification) or 50 % if ischemia corresponding to the target lesion is documented either by exercise stress ECG, stress echocardiography, scintigraphy, MRT, or suspected based on angina pectoris
* Single or multi-vessel coronary artery disease

Exclusion Criteria:

Patient Exclusion Criteria

* Exclusion Criteria: Patient Related
* Patients with acute (<24 h) or recent (48 hours) myocardial infarction
* Patients with unstable angina pectoris (Braunwald class 3)
* Patients with severe congestive heart failure
* Patients with severe heart failure NYHA IV
* Patients demonstrating clinical signs of cardiogenic shock at the time of the procedure (systolic blood pressure of less than 80 mmHg requiring inotropic support, IABP, and/or fluid challenge)
* Patients with severe valvular heart disease
* Women who are pregnant or lactating
* Patients with life expectancy of less than five years or factors making clinical follow-up difficult
* Patients with bleeding diathesis in whom anticoagulation or anti-platelet medication is contraindicated
* Patients who had a cerebral stroke <6 months prior to the procedure
* Patient participates in other clinical trials involving any investigational device or drug
* Untreated hyperthyroidism
* Patient has presence or history of severe renal failure (GFR<30ml/min, "Cockcroft Gault") and is therefore at high risk for angiography associated renal complications. Patient's serum creatinine levels must be documented
* Post transplantation of any organ or immune suppressive medication
* Other disease to jeopardize follow-up (e.g,malignancy)
* Addiction to any drug or to alcohol
* Patients with any type of surgery during the week preceding the interventional procedure.
* Therapy with anticoagulants
* After PTCA,Coronary artery dissection appears Exclusion Criteria: Lesion Related
* Evidence of extensive thrombosis within target vessel before the intervention
* Multilesion percutaneous coronary intervention beside the bifurcation lesion in the left coronary artery (no other intervention is admitted during the same procedure)
* Patients with another coronary stent implanted previously into the target vessel ≤15 mm distant to the current lesion, drug eluting stents less than 9 months and bare metal stents or stents with passive coatings less than 3 months before the PEBCBLO
* Target lesion located in any type of coronary bypass (i.e,venous graft, arterial bypass) or graft/native artery connection
* Coronary artery occlusion of any type (e.g, acute or chronic)
* In-stent restenosis
* In-segment restenosis of the native vessel within 4 mm adjacent to the target lesion Exclusion Criteria Related to Concomitant Medication
* Patient is intolerant to aspirin and/or the ADP-antagonists clopidogrel/ticlopidine or has a history of neutropenia, thrombocytopenia induced by ADP-antagonists, or severe hepatic dysfunction prohibiting the use of clopidogrel

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is designed for 25 subsequent patients with coronary heart disease to complete the study per protocol. Eligible patients shall exhibit a bifurcational lesion in the native left coronary artery (reference diameter LAD or LCx: 2.5 mm -4.0 mm, length of stenosis: ≤30 mm, reference diameter D1/D2 or OMS1/OMS2: 2.0 mm-3.5 mm, length of stenosis: ≤ 30 mm) in need of percutaneous coronary intervention. Eligible patients may have single or multivessel coronary artery disease.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-01 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
In-segment late lumen loss | 9 months
  In-segment late lumen loss in the side branch and main branch evaluated by OCT

SECONDARY OUTCOMES:
major adverse cardiac events (MACE) | 9 months
  cardiac death, myocardial infarction and target lesion revascularization
Procedural success | 10 minutes
  a stenosis ≤30% in the MB and ≤50% in the SB along with TIMI III flow

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Jilin University, Changchun, Jilin, China